CLINICAL TRIAL: NCT01746602
Title: Effect of Topical Glaucoma Therapy on Tear Film Stability in Healthy Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-241010
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: topical lubricants; tear film thickness; anti-glaucoma drugs; break up time; anti-glaucoma treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- healthy subjects I (Experimental): 20 healthy subjects
  Interventions: Drug: Timoptic® 0.5%
- healthy subjects II (Experimental): 20 healthy subjects
  Interventions: Drug: Timophtal sine® 0.5%
- healthy subjects III (Experimental): 20 healthy subjects
  Interventions: Device: Genteal HA®
- healthy subjects IV (Experimental): 20 healthy subjects
  Interventions: Device: Hylo-Comod®
- healthy subjects V (Experimental): 20 healthy subjects
  Interventions: Device: Thealoz®
- healthy subjects VI (No Intervention): 20 healthy subjects

INTERVENTIONS:
Drug: Timoptic® 0.5% — Timoptic® 0.5% Eye Drops, Merck, single instillation
  Arms: healthy subjects I
Drug: Timophtal sine® 0.5% — Timophtal sine® 0.5%, Agepha, Eye Drops, single instillation
  Arms: healthy subjects II
Device: Genteal HA® — Genteal HA® Eye Drops, Novartis, single instillation
  Arms: healthy subjects III
Device: Hylo-Comod® — Hylo-Comod® Eye Drops, Croma-Pharma, single instillation
  Arms: healthy subjects IV
Device: Thealoz® — Thealoz® Eye Drops, Thea, France, single instillation
  Arms: healthy subjects V

SUMMARY:
Long term treatment with anti-glaucomatous drugs has been shown to increase the incidence of dry eye syndrome with all known consequences such as ocular discomfort and epithelial keratitis. Given that thinning of the tear film appears to be a risk factor for the development or the aggravation of dry eye syndrome, the current study seeks to investigate whether tear film thickness is changed after topical treatment with anti-glaucomatous drugs in healthy subjects.

For this purpose, tear film thickness will be measured at baseline and after single instillation of one of 5 study drugs in one randomly chosen eye. In addition, one group of 20 subjects will receive no drug and will serve as a second control. Drug effects on tear film thickness will be compared to the fellow, non-treated eye. In addition, effects on tear film thickness of timolol with preservatives (Timoptic 0.5%) will be compared to timolol without preservatives (Timophtal sine 0.5%) and three lubricants with different viscosity (Genteal HA, Hylo-Comod, Thealoz).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt.

Exclusion Criteria:

* Regular use of medication (except contraceptives), abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Patients with known hypersensitivity to the study drug or any ingredients
* History or current COPD or asthma
* AV-block grade II or more
* Ametropy ≥ 6 Dpt
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Tear film thickness | up to 1 hour

SECONDARY OUTCOMES:
Break up time (BUT) | once on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Werkmeister RM, Alex A, Kaya S, Unterhuber A, Hofer B, Riedl J, Bronhagl M, Vietauer M, Schmidl D, Schmoll T, Garhofer G, Drexler W, Leitgeb RA, Groeschl M, Schmetterer L. Measurement of tear film thickness using ultrahigh-resolution optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 Aug 15;54(8):5578-83. doi: 10.1167/iovs.13-11920. PMID 23847319